CLINICAL TRIAL: NCT03136549
Title: Cuff Inflation-supplemented Videoscope-guided Nasal Intubation: The Effect of Tube Thermo-softening on the Nasotracheal Navigability
Brief Title: Cuff Inflation-supplemented Videoscope-guided Nasal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jun joohyun, assistant professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-03-020
Record Dates: First submitted 2017-04-19; First posted 2017-05-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Nasotracheal Intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Room temperature (Placebo Comparator): The nasotracheal tube, sized 6.0 -7.0 mm inner diameter (ID), were put into a bottle of sterilized normal saline (1 L, 25 °C) at room temperature.
  Interventions: Other: Room temperature
- Thermo-softening (Experimental): The naso tracheal tube, sized 6.0 -7.0 mm inner diameter (ID), were put into a bottle of sterilized normal saline (1 L) at warm cabinet set to 45°C (approximately 117°F).
  Interventions: Other: Thermo-softening

INTERVENTIONS:
Other: Thermo-softening — The thermosoftening treatment of the tubes was performed by using a warm cabinet set to 45°C (approximately 117°F). One bottle of normal saline (1 L) containing a thermometer and three tubes (6.0 -7.0 mm ID) was put into a chamber of the cabinet 30 min before intubation.
  Arms: Thermo-softening
Other: Room temperature — nasotracheal tube, sized 6.0 -7.0 mm inner diameter (ID), were put into a bottle of sterilized normal saline (1 L, 25 °C) at room temperature.
  Arms: Room temperature

SUMMARY:
Epistaxis or post-pharyngeal bleeding is the most common complication after nasotracheal intubation (NTI). Prior thermal softening of the endotracheal tube (ET) has been recommended as one of the methods to prevent nasal trauma from nasotracheal intubation. However, thermal softening of tubes tends to adversely affect the nasotracheal navigation of the ET.

During NTI under conventional direct laryngoscopy, the tip of the Macintosh laryngoscope is advanced into the vallecula, indirectly elevating the epiglottis by applying pressure on the hyoepiglottic ligament. Although this maneuver allows optimal visualization of the glottis, it lifts the larynx away from the tip of the advancing nasotracheal tube (NTT), which generally lies along the posterior pharyngeal wall. Most clinicians use Magill forceps to direct the tip of the NTT anteriorly to enter the glottis. Magill forceps may cause damage to the cuff of an ET or may injure oropharyngeal mucosa.

The use of a video laryngoscope and a cuff inflation technique has been proposed as a method for reducing the malalignment of tubes. Indirect laryngoscopy using a Video laryngoscopy can reduce malalignment by minimizing lifting the glottis during laryngoscopy. The cuff inflation technique (wherein the cuff of ET tube is inflated with 15 mL of air) has been used while performing "blind" NTI to guide such malaligned polyvinyl chloride (PVC) ET tubes into the laryngeal inlet. Recently, one study reported that the cuff inflation technique consistently improved the oropharyngeal insertion of the different ET tubes of varying stiffness during direct laryngoscope-guided NTI.

There has never been study about effect of cuff inflation technique on navigability when performing NTI under video laryngoscopy guidance with ET tubes of varying stiffness.Investigators assessed and compared the incidence of nasal injury and nasotracheal navigability with two technique during cuff inflation-supplemented NTI guided by video- laryngoscopy

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-III, older than 18 yr, who under went elective surgery and requiring ET intubation as part of anesthetic management were enrolled in the study.

Exclusion Criteria:

* Patients with bleeding diathesis, history of recurrent nasal obstruction or any nasal/pharyngeal surgery, and those with anticipated difficult tracheal intubation were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
severity of epistaxis | during navigation from nose to oropharynx
  The severity of epistaxis was evaluated under VL using a 4-point scale:no epistaxis; mild epistaxis (blood on the tracheal tube only); moderate epistaxis (blood pooling in the pharynx); or severe epistaxis (blood in the pharynx sufficient to impede intubation)

SECONDARY OUTCOMES:
the navigation of ET tube from nose to oropharynx | during navigation from nose to oropharynx
  The navigability (ease of insertion) was scored as grade 1 if the tube advanced smoothly from the nose into oropharynx, grade 2 if there was resistance in the passage that could be managed by side-to-side rotation of the tube, and grade 3 if the tube impinged unduly and the other nostril had to be used.
time | The passage of each ET tube from nasal cavity to trachea was divided into 3 phases (phase 1: from the nose into oropharynx, phase 2: from oropharynx into the laryngeal inlet , phase 3: from the laryngeal inlet into the trachea)
  time required for passage of tube in each phase
air volume | during navigation from oropharynx to laryngeal inlet
  the volume of air needed for cuff inflation during navigation from oropharynx to laryngeal inlet
the navigation of ET tube from oropharynx to laryngeal inlet | during navigation from oropharynx to the laryngeal inlet
  The tube was then advanced further from oropharynx into the laryngeal inlet under video laryngoscopic vision, and a smooth passage was scored as grade 1. In case the tube failed to align with the laryngeal inlet, the tube tip was withdrawn into the laryngopharynx and the cuff of the tube was sequentially inflated with air in 4 mL aliquots up to a maximal volume of 40 mL by an assistant on request until it aligned with the laryngeal inlet (cuff inflation technique) and got engaged in it thereafter (grade 2). If this technique was unsuccessful, the cuff was deflated and Magill forceps were used to engage the tube tip into the laryngeal inlet (grade 3).
the navigation of ET tube from laryngeal inlet to trachea | during navigation from laryngeal inlet to trachea
  A smooth passage was considered grade 1. If the ET tube tip got stuck in the laryngeal vestibule, optimal external laryngeal manipulation (OELM) applied (grade2); If the ET tube tip got stuck in the laryngeal vestibule, it was rotated clockwise while maintaining a gentle forward pressure on it until it got disengaged from its impingement and then slipped into the trachea (grade 3). In case this maneuver was unsuccessful, Magill forceps were used to complete the intubation process (grade 4).

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No